CLINICAL TRIAL: NCT06282744
Title: Cross Cultural Adaptation, Validity and Reliability Test of the Arabic Version of the Outpatient Physical Therapy Improvement in Movement Assessment Log
Acronym: OPTIMAL
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Hamdy Abdeltwab Hussien, Dr Eman Hamdy, Cairo University
Other Study IDs: OPTIMAL Arabic version
Record Dates: First submitted 2024-01-14; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Physical Performance; Outpatients
Keywords: Questionnaire; OPTIMAL; Validity testing; Arabic version; Psychometric properties; Reliability Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Outpatient physical therapy improvement in movement assessment log — The Outpatient Physical Therapy Improvement in Movement Assessment Log (OPTIMAL) is an instrument that measures difficulty and self-confidence in performing 22 movements that a patient needs to accomplish in order to do various functional activities.

SUMMARY:
Purpose of the study:

To translate, culturally adapt, and to test the validity and reliability of the Outpatient Physical Therapy Improvement in Movement Assessment Log in Arabic speaking language.

DETAILED DESCRIPTION:
The OPTIMAL assessment log was produced in English and later on it was being validated into Italian and Spanish versions. It hasn't been produced into Arabic yet so the aim of this study is to test the validity , reliability and psychometric properties of this assessment tool when being translated into Arabic and used among the Arabic Egyptian people.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are adult outpatients who took at least a month of physiotherapy sessions.
2. Both genders will be included.
3. At least 18 years of age.
4. Participants must be conscious and ambulant.
5. Participants able to read, write Arabic as a mother tongue and understand the instructions, questions in the questionnaire.

Exclusion Criteria:

Participants having the following conditions will be excluded from the study:

1. Patients who are not able to provide informed consent.
2. Patients who are unable to complete the OPTIMAL instrument.
3. Patients who have a severe cognitive impairment.
4. Patients who are not receiving physical therapy.
5. Patients who are not Arabic-speaking.
6. Patients who have a history of malingering

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Egyptian adults who took at least a month of physiotherapy sessions.
Sampling Method: Non-Probability Sample
Enrollment: 880 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
validity and reliability of the Egyptian Arabic language version of Outpatient Physical Therapy Improvement Movement Assessment Log on physical therapy outpatients. | Up to 24 weeks
  to test if the Arabic version of this log is valid for usage among Egyptian People. Test improvement in different movements.